CLINICAL TRIAL: NCT04188028
Title: Endobiotics for Phenotyping of Human Cytochrome P450 Enzymes: Use of Metabolomics for the Identification of New CYP2D6 Endogenous Biomarkers in Healthy Volunteers
Brief Title: Endobiotics for Phenotyping of Human Cytochrome P450 Enzymes
Acronym: ENDOCYP2D6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-01637
Record Dates: First submitted 2019-04-18; First posted 2019-12-05 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dextromethorphan; Paroxetine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYP2D6 gene score 0 (Experimental): CYP2D6 gene score 0: carrier of two non-functional alleles
  Interventions: Drug: Dextromethorphan 5 MG; Drug: Paroxetine 10Mg Tablet
- CYP2D6 gene score ≥1 (Experimental): CYP2D6 gene score ≥1: carrier of one fully-functional and one non-functional allele of CYP2D6 , one fully-functional and one reduced-function of CYP2D6, two fully-functional alleles of CYP2D6 or more than two functional alleles alleles
  Interventions: Drug: Dextromethorphan 5 MG; Drug: Paroxetine 20Mg Tablet

INTERVENTIONS:
Drug: Dextromethorphan 5 MG — dextromethorphan 5 mg po
Drug: Paroxetine 10Mg Tablet — Paroxetine 10 mg po
  Arms: CYP2D6 gene score 0
Drug: Paroxetine 20Mg Tablet — Paroxetine 20 mg po
  Arms: CYP2D6 gene score ≥1

SUMMARY:
CYP2D6 metabolizes ~25% of all marketed drugs. There is an important variability in the activity of this enzyme among individuals. The cause of this variability might be environmental, genetic, ethnical or even related to a disease. The administration of a CYP2D6 probe drug (e.g. dextromethorphan) is a good way to characterize CYP2D6 phenotype. Nonetheless, it is relatively invasive and the vulnerable population (e.g. pregnant women) cannot be phenotyped in this manner. Therefore, finding an endogenous substance which is metabolized by CYP2D6 could replace usual phenotyping procedure using a probe drug. This study evaluates the impact of a CYP2D6 inhibitor and of genetic polymorphism on the metabolome of healthy volunteers in order to identify new CYP2D6 biomarkers. To this end, untargeted metabolomics analysis using LC-HRMS will be performed on plasma and urine samples This single-centre open-label clinical trial will include 40 healthy subjects (men and women) between 18 and 65 years. Eligible participants will be assigned to a study group according to their CYP2D6 genotypes: poor metabolizers (PMs) and extensive/ultrarapid metabolizers (EMs-UMs). Two sessions will take place for each subjects.

Session 1: CYP2D6 phenotyping (dextromethorphan 5 mg, single dose) Session 2: idem session 1 with prior uptake of a CYP2D6 inhibitor (paroxetine 10 or 20 mg, one dose a day for 7 days).

In both sessions, urine will be collected up to 24 hours and capillary/venous blood will be sampled before phenotyping for metabolomics analyses. Urine will also be collected for 4 hours after dextromethorphan intake in order to phenotype the CYP2D6 enzyme.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-65 years
* Body Mass Index (BMI) 18-27
* Understanding of French language and able to give a written inform consent
* CYP2D6 genotype : activity score = 0 (PMs) or activity score ≥ 1 (EMs-UMs)
* Reliable contraception during the whole study, including a barrier method

Exclusion Criteria:

* Participation in any other interventional clinical study within 3 months prior to inclusion
* Pregnant or breastfeeding woman
* Any pathologies, use of drugs or food that may affect CYP activity (based on the 'drug interactions and cytochromes P450' table published by the Service of Clinical Pharmacology and Toxicology, HUG54 and on the investigator's knowledge)
* Regular smokers of ≥ 10 cigarettes/day
* Alcohol intake 2 days prior to session 1 and during paroxetine intake
* Medical history of chronic alcoholism or abuse of psychoactive drugs
* Regular use of psychotropic substances
* Sensitivity to any of the drugs used
* Alteration of hepatic tests (ASAT, ALAT, BILI, GGT) more than 3x normal
* Psychiatric disorders
* Beck Score ≥10 (question related to suicide >0)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Identify endogenous markers of CYP2D6 activity in urine and plasma using untargeted metabolomics | 7 days
  Metabolomic strategie (LC-Q-Exactive HRMS) will be used to identify and characterize endogenous compounds that correlate with the urinary metabolic ratio dextromethorphan/dextrorphan before and after administration of paroxetine, a strong CYP2D6 inhibitor.

SECONDARY OUTCOMES:
Difference in DEM/DOR urinary ratio before and after administration of paroxetine | 7 days
Correlation of significant ions with DEM/DOR urinary ratio or CYP2D6 activity score | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided